CLINICAL TRIAL: NCT06221553
Title: Safety and Efficacy of Intraventricular Infusion of B7H3 With IL-7 Receptor Alpha Signaling Chimeric Antigen Receptor T Cell in Diffuse Intrinsic Pontine Glioma
Brief Title: Safety and Efficacy of Loco-regional B7H3 IL-7Ra CAR T Cell in DIPG
Acronym: CMD03DIPG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LV-B7H3IL7-CART-DPG-P1-2023; Chulalongkorn University (Other: Chulalongkorn University)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: DIPG Brain Tumor; Diffuse Intrinsic Pontine Glioma
Keywords: CAR T cell; DIPG; B7H3; IL-7 receptor alpha; Chimeric antigen receptor T cell; Adoptive cellular therapy
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locoregional delivery of B7H3/IL-7Ra CAR T cell in DIPG (Experimental): Patients with DIPG for whom CAR T cells will be delivered into the ventricular system
  Interventions:
  Biological: Autologous B7H3-specific chimeric antigen receptor (CAR) T cell with additional of IL-7Ra signaling domain Dose level: 1x10e7 CAR T cell, 3x10e7 CAR T cell, 10x10e7 CAR T cell
  Interventions: Biological: B7H3 specific CAR T cell with IL-7Ra signaling domain

INTERVENTIONS:
Biological: B7H3 specific CAR T cell with IL-7Ra signaling domain — Autologous T cells lentivirally transduced to express a B7H3 specific chimeric antigen receptor (CAR) with additional of IL-7 receptor alpha signalingdomain given via indwelling central nervous system (CNS) catheter

SUMMARY:
A Phase 1 clinical trial to evaluate the safety and early efficacy of CAR T-cell with IL-7Ra signal targeting B7H3 in children with diffuse intrinsic pontine glioma (DIPG) patients after complete standard treatments.

DETAILED DESCRIPTION:
The brain tumor known as Diffuse Intrinsic Pontine Glioma is commonly found in children aged between 5 to 10 years. This type of tumor is aggressive and infiltrates the structures of the brain stem. Treatment options are limited due to the location of the tumor, making it impossible to surgically remove the mass like other brain cancers. The standard treatment for this type of tumor is radiation therapy, as this type of cancer does not respond to chemotherapy or currently available targeted drugs. However, radiation therapy has been found to be ineffective and does not improve survival rates.

Currently, there is development in cancer treatment using immunotherapy, where the patient's immune cells are genetically modified to target the cancer, also known as CAR T cells, for the treatment of recurrent or refractory cancers in solid tumors and brain cancers. The research project aims to study the efficacy and safety of treating patients with pontine glioma using T cells that are antigen-specific and have signals from the interleukin-7 receptor alpha and are specific to the B7H3 antigen on the tumor surface. This research is the first of its kind in Thai patients. The research project expects that this treatment will be highly safe and effective in controlling diffuse pontine glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have diffuse intrinsic pontine glioma at any timepoint following completion of standard radiotherapy
2. Age 1-18 years
3. Sex: Male or female
4. CNS reservoir catheter, such as an Ommaya or Rickham catheter, present in the proper location for CNS-directed therapy
5. Performance status: Lansky or Karnofsky score >= 60
6. Life expectancy >= 8 weeks
7. Normal organ function:

   7.1 AST (SGOT) < 5 times the upper limit of normal (ULN) 7.2 ALT (SGPT) < 5 times the upper limit of normal (ULN) 7.3 Total bilirubin < 3 times the upper limit of normal (ULN) 7.4 Creatinine < 5 times the upper limit of normal (ULN) 7.5 SpO2 room air >=90%
8. Prior therapy wash-out before planned leukapheresis 8.1 >= 7 days post last chemotherapy/biologic therapy administration 8.2 3 half-lives or 30 days, whichever is shorter after the last dose of antitumor antibody therapy 8.3 At least 30 days from most recent cellular infusion 8.4 All systemically administered corticosteroid treatment therapy must be stable or decreasing within 1 week prior to enrollment with a maximum dexamethasone dose of 2.5 mg/m2/day. Corticosteroid physiologic replacement therapy is allowed
9. Participants and/or legal guardians must have the ability to understand and willingness to sign a written informed consent and/or assent document

Exclusion Criteria:

1. Presence of >= grade 3 cardiac dysfunction or symptomatic arrythmia requiring intervention
2. Presence of primary immunodeficiency or bone marrow failure syndrome
3. Presence of clinical and/or radiographic evidence of impending herniation of CNS
4. Presence of > Grade 3 dysphagia
5. History of active malignancy other than nonmelanoma skin cancer and carcinoma in situ (e.g., cervix, bladder, breast).
6. Presence of uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant or breastfeeding women were excluded from this study because CAR-T-cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study. Participants of childbearing or child-fathering potential must be willing to practice birth control from the time of enrollment in this study and for four months after receiving CAR-T-cell infusion.
8. Serologic status reflecting active HIV, hepatitis B or C infection. Participants who are positive for hepatitis B core antibody, hepatitis B surface antigen or hepatitis C antibody must have negative PCR prior to enrollment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety of B7H3-IL7Ra CAR T cells infusion in diffuse intrinsic pontine glioma (DIPE) patients. | Up to 28 days after B7H3-IL7Ra CAR-T cell infusion
  The incidence of adverse events assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0

SECONDARY OUTCOMES:
The overall response rate of diffuse intrinsic pontine glioma (DIPE) | 3, 6, and 12 months after B7H3-IL7Ra CAR-T cell infusion
  The overall response rate will be assessed using radiologic response criteria that use the standard sum of the two longest 2D perpendicular diameters to distinguish stable disease, progressive disease (>25% increase), partial response (>50% decrease), and complete response (no evaluable or measurable disease).

OTHER OUTCOMES:
The persistence and distribution of B7H3-IL7Ra CAR T cells in the CSF and peripheral blood | 14 days, 28 days, 42 days 3 months, 6 months, and 12 months after B7H3-IL7Ra CAR-T cell infusion
  The persistence and distribution of B7H3-IL7Ra CAR T cells in the CSF and peripheral blood of diffuse intrinsic pontine glioma patients will be measured by flow cytometry.
Serum cytokine level measurement | 1 day, 14 days, 28 days and 42 days after B7H3-IL7Ra CAR-T cell infusion.
  Serum cytokine level measurement before and after B7-H3-IL7Ra CAR T-cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Piti Techavichit, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No